CLINICAL TRIAL: NCT03682627
Title: PREventive Effect of FENestration With and Without Clipping on Post-Kidney Transplantation Lymphatic Complications: PREFEN Trial
Brief Title: Preventive Fenestration With and Without Clipping in Kidney Transplantation
Acronym: PREFEN
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University Hospital Heidelberg (Other)
Responsible Party: Principal Investigator, Dr. A. Mehrabi, Professor Dr. med., University Hospital Heidelberg
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: S-318/2017
Record Dates: First submitted 2018-09-18; First posted 2018-09-24 (Actual); Last update posted 2018-09-24 (Actual); Status verified 2018-09

CONDITIONS: Kidney Transplantation
Keywords: kidney transplantation; Lymphatic complications; preventive fenestration; clipping
MeSH Terms: interventions — Fenestration, Labyrinth

STUDY DESIGN:
Intervention Model Description: single intuition, double blinded, randomized clinical trial.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- preventive fenestration (Active Comparator): Fenestration is performed at the time of kidney transplantation
  Interventions: Procedure: Fenestration
- preventive fenestration and clipping (Experimental): Fenestration and clipping of the edges are performed at the time of kidney transplantation
  Interventions: Procedure: Fenestration and clipping

INTERVENTIONS:
Procedure: Fenestration — A standardized fenestration of the peritoneum will be performed. A 2 cm incision will be made in the peritoneum that is parallel to the skin incision after the transplant procedure. The peritoneal will not be sutured at the edges to keep the fenestration open. No interpositioning of the omentum will be performed.
  Arms: preventive fenestration
Procedure: Fenestration and clipping — A standardized fenestration of the peritoneum will be performed. A 2 cm incision will be made in the peritoneum that is parallel to the skin incision after the transplant procedure. The window edges will be clipped after fenestration using 8 metal clips.
  Arms: preventive fenestration and clipping

SUMMARY:
Post-Kidney Transplantation Lymphatic complications include lymphorrhea and lymphocele, and are some of the most challenging issues after kidney transplantation. The most frequent post-Kidney transplantation complication is accumulation of perirenal fluids, such as urinomas, hematomas, and lymphoceles. Lymphoceles are associated with morbidities such as abdominal discomfort, impaired wound healing, and thrombosis. Lymphoceles may also affect graft function by putting direct pressure on the kidney, or by compressing the ureter or transplant vasculature. The frequency and consequences of post-transplantation lymphoceles make preventive measures highly desirable. Peritoneal fenestration during kidney Transplantation is a simple method for preventing lymphocele formation. Recent studies have evaluated the effectiveness of clipping with metallic clips following fenestration on lymphocele formation and lymph leakage after prostate cancer surgery and laparoscopic retroperitoneal lymph node dissection. However, whether clipping prevents lymphocele formation after kidney transplantation has not been investigated. The aim of the proposed study is to compare the effect of fenestration with and without clipping on incidence of post-kidney transplantation lymphocele and lymphorrhea.

DETAILED DESCRIPTION:
Recent improvements in transplantation techniques, organ matching systems, and modern immunosuppressive regiments have made kidney transplantation a routine operation with acceptable mortality and morbidity rates. Post-kidney transplantation morbidities include vascular and urological complications, and postoperative fluid collections. Perirenal fluid collections, such as urinomas, hematomas, and lymphoceles, are some of most frequent complications following Kidney transplantation, among which post-Kidney transplantation lymphatic collections, are most challenging complications.

The incidence of post-kidney transplantation lymphatic complications is up to 50% and the peak incidence of lymphocele is during the 6th postoperative week (range: 2 weeks to 6 months).

Lymphoceles are usually asymptomatic and identified incidentally by routine ultrasound examination. However lymphoceles may result in morbidities such as abdominal discomfort, impaired wound healing, and thrombosis. Post-kidney transplantation lymphatic complications may also affect graft function by putting pressure on the kidney, or by compressing the ureter or transplant vasculature. The frequency and consequences of post-transplantation lymphoceles make preventive measures highly desirable.

Various preventive methods have been proposed in the literature. Lymphoceles usually originate from unligated lymphatic vessels, therefore precise ligation of donor and recipient lymphatic vessels can reduce lymphocele formation. Compression therapy of the lower limb after kidney transplantation and appropriate immunosuppressive therapy may also reduce lymphocele formation. Some authors have used polymeric sealants/hemostatic biomaterials or povidone-iodine to prevent lymphocele formation. However, the effectiveness and cost-efficiency of these methods has not been conclusively proven. Use of drains in lymphocele prevention has also been previously suggested, but this method remains controversial. Peritoneal fenestration at the time of kidney transplantation is a simple method to prevent lymphocele formation. This method has been widely studied in treatment and prevention of lymphoceles following kidney transplantation. However, to the best of our knowledge, only one randomized controlled trial has been performed to investigate the impact of preventive fenestration in prevention of post kidney transplantation lymphatic complications. This study showed that the prevalence of fluid collections in the fifth postoperative week was significantly higher in the standard group compared to fenestration group. Also, 15.5% of patients in the standard group developed symptomatic lymphoceles requiring treatment during the first postoperative year, versus 3.0% in the fenestration group.

Recent studies have evaluated the effectiveness of extensive clipping using metallic clips following fenestration on lymphocele formation and lymph leakage after prostate cancer surgery and laparoscopic retroperitoneal lymph node dissection. Some surgeons have declared concerns that larger fenestrations increase the risk of hernia. However, risk of closure of the peritoneal fenestration is higher for smaller Windows in the peritoneal cavity. Recently clipping of the edges of peritoneal fenestration was performed in the surgical clinic of the Heidelberg University Hospital to reduce risk of closure of the fenestration after kidney transplantation. However, whether fenestration and clipping prevents lymphocele formation after kidney transplantation has not been investigated.

This clinical Trial is designed to investige the rate of post-kidney transplantation lymphocele and lymphorrhea in two groups of kidney transplantation patients: one with only fenestration and one with fenestration and clipping of the edges. Additionally, graft function and incidence rate of other morbidities will be investigated and analyzed after transplantation.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Provide written informed consent
* Recipients of KTx from deceased donors

Exclusion Criteria:

* Inability to comply with study and/or follow-up procedures
* Recipients of KTx from living donors
* Combined transplantation (e.g. pancreas-kidney transplantation)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Estimated)
Dates: Start 2018-10 (Estimated); Primary Completion 2020-09 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Post kidney transplantation lymphocele | 6 months
  Fluid collection of variable size located near to the transplanted kidney in a non-epithelialized cavity. The possibility that the accumulation of fluid is a hematoma, abscess, and urinoma will be ruled out after aspiration of the fluid.

SECONDARY OUTCOMES:
Operation time | 1 day
  From skin incision to skin closure
Estimated blood loss | 1 day
  Blood loss during operation from skin incision to skin closure (mL)
Length of hospital stay | 6 months
  From the time of the operation to time of discharge
Postoperative complications | 6 months
  Postoperative complications will be reported and classified according to the Clavien-Dindo classification.
Mortality | 90 days
  Death due to any cause.
Post Kidney transplantation fluid collection | 6 months
  Fluid accumulation near to the transplanted kidney will be diagnosed by ultrasound as routine of the Heidelberg
Post Kidney transplantation lymphorrhea | 6 months
  Defined as an outflow of more than 50 (milileter) of fluid per day after the 7th post-KTx day. Fluid that flows from the drain, or the site of the removed drain, or surgical wound, which is not blood, pus, or urine will be monitored
Lymphocele size | 6 months
  Lymphocele diameter and volume will be recorded by ultrasound examination in mL.
Lymphocele symptomes | 6 months
Lymphocele/lymphorrhea severity grade | 6 months
  Severity of lymphocele/lymphorrhea will be graded based on the applied management strategy (Grade A: Observation, Grade B: Non-surgical intervention, Grade C: Surgery).
Blood Urea Nitrogen Level | 6 months
  Blood Urea Nitrogen Level (mg/dL)
Plasma uric acid Level | 6 months
  Plasma uric acid Level (mg/dL)
Serum creatinine level | 6 months
  Serum creatinine level (mg/dL)
Rate of delayed graft function | 30 days
  Is defined as the need for one or more hemodialysis treatments following transplantation prior to the onset of graft function.
Glomerular filtration rate | 6 months
  GFR (mL/min/1.73 m2) calculated with "175 × (Scr)-1.154 × (Age)-0.203 × (0.742 if female)" Formula
Rate of primary non-function grafts | 30 days
  number of recipients whose grafts never functions after transplantation
Retransplantion rate | 6 months
  Rate of retransplantation

CONTACTS AND LOCATIONS:
Overall Officials: Arianeb Mehrabi, MD, Principal Investigator — Department of General, Visceral and Transplant Surgery, University Hospital
Locations (1):
- Division of Visceral Transplantation, Department of General, Visceral and Transplantation Surgery, University of Heidelberg, Heidelberg, Baden-Wurttemberg, Germany

REFERENCES:
- [Derived] Golriz M, Sabagh M, Mohammadi S, Ghamarnejad O, Khajeh E, Mieth M, Al-Saeedi M, Diener MK, Mihaljevic AL, Morath C, Zeier M, Kulu Y, Mehrabi A. PREventive effect of FENestration with and without clipping on post-kidney transplantation lymphatic complications (PREFEN): study protocol for a randomised controlled trial. BMJ Open. 2020 Oct 13;10(10):e032286. doi: 10.1136/bmjopen-2019-032286. PMID 33051226